CLINICAL TRIAL: NCT06018051
Title: Evaluation of the Concept "Can Do" Versus "Do Do" in Patients With Breast Cancer
Brief Title: "Can Do" Versus "Do Do" in Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Associate Professor, Hacettepe University
Other Study IDs: GO 23/582
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Exercise Capacity; Physical Activity
Keywords: breast cancer; Quality of life.; exercise; physical activity; Physical capacity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer occurs as a result of uncontrolled proliferation of cells in the breast tissue. Breast cancer is the most common type of cancer among women worldwide and is an important problem that threatens women's lives. The incidence rate has reached approximately 16 Breast cancer treatment consists of local and systemic therapies. While local treatments include surgery and radiotherapy, systemic treatments, which are administered in two different ways, namely adjuvant and neoadjuvant systemic treatments, consist of chemotherapy, hormone therapy and targeted biological therapies. Although the treatment options for breast cancer are increasing day by day, there are many complications during and after treatment. These complications negatively affect functionality and quality of life The 6-minute walk test (6MWD) is a widely used test for indirect measurement of cardiorespiratory fitness in various cancer populations. Studies have proven that the 6MWT is safe and feasible in breast cancer patients. The concept of 'can do, do do' has recently emerged to describe impaired physical functions in chronic obstructive pulmonary disease (COPD) and asthma. This concept categorizes participants into four quadrants based on physical activity level and functional capacity measurements and cut-off point. This concept has proven useful for measuring physical function in both asthma and COPD. This concept may be useful in understanding physical functioning in breast cancer patients. Therefore, The aim of this study is to apply the concept of 'can do, do do' in breast cancer patients, to determine the quadrants according to physical activity level and functional capacity measurements in breast cancer patients, to investigate whether and to what extent there is a difference, whether and to what extent there is a difference between demographic information, disease stages, comorbidity level, clinical features, peripheral muscle strength, fatigue and quality of life and upper extremity functionality according to quadrants.

DETAILED DESCRIPTION:
Breast cancer occurs as a result of uncontrolled proliferation of cells in the breast tissue. Breast cancer is the most common type of cancer among women worldwide and is an important problem that threatens women's lives. The incidence rate has reached approximately 16 Breast cancer treatment consists of local and systemic therapies. While local treatments include surgery and radiotherapy, systemic treatments, which are administered in two different ways, namely adjuvant and neoadjuvant systemic treatments, consist of chemotherapy, hormone therapy and targeted biological therapies. Although the treatment options for breast cancer are increasing day by day, there are many complications during and after treatment. These complications negatively affect functionality and quality of life.

Thanks to the increasing treatment possibilities with the developing technology in recent years, the majority of patients show good functional recovery after breast cancer. However, it has been reported that treatments negatively affect the functional capacity of the upper extremities, daily life, work and social activities and decrease the quality of life. Many side effects are observed in patients after breast cancer treatment. Therefore, there are various rehabilitation needs. Side effects vary from person to person. Therefore, the rehabilitation program to be applied should be personalized. Commonly reported side effects of the disease or treatments include pain, lymphedema, fatigue and depression. In addition, psychosocial consequences and psychological distress, such as reduced health-related quality of life and reduced social contacts, as well as difficulties in maintaining functional activities and life roles, have been reported. As a result, breast cancer patients may have physical, psychological, social and existential rehabilitation needs.

Exercise is an effective non-pharmacologic treatment method in cancer patients. Exercise also has therapeutic properties in cancer-related fatigue. Increased physical activity has been reported to improve psychological recovery and physical well-being in cancer patients. Aerobic exercise has been proven to reduce cancer-related fatigue as a result of studies. It has also been reported that supervised exercise during chemotherapy or radiotherapy treatments both increases the effectiveness of the treatment and reduces the side effects that may occur. In addition, resistance exercises significantly reduce cancer-related fatigue. There is evidence that there is a strong relationship between the risk of breast cancer and physical activity level. Exercise training is an important physiotherapy and rehabilitation approach in breast cancer survivors. According to randomized controlled trials on the outcomes of exercise modalities in women with breast cancer, women who exercise have improved survival rates. Physical and psychological conditions such as fatigue, pain, anxiety, depression and decreased functional capacity reduce patients' quality of life. Exercise interventions during or after treatment have been reported to improve musculoskeletal performance, cardiorespiratory fitness, body awareness, and psychological status in breast cancer. Previous studies have also reported that exercise training programs to be applied during or after cancer treatment in cancer patients improve quality of life. It has been reported that mind-body togetherness exercises such as aerobic, resistance, stretching, yoga, and Tai Chi in breast cancer patients improve quality of life and general and mental health, and have a positive effect on of the maximal oxygen uptake (VO2 max) , and provide significant improvements in self-esteem and attitude towards life. In addition, exercise training alleviates symptoms of depression and anxiety in breast cancer survivors. In addition to reducing body mass index (BMI) and causing significant increases in lean mass, exercise also increases muscle strength in the intervention groups. Furthermore, the serum concentration of some physiological markers, such as insulin, insulin-like growth factor (IGF-II) and insulin-like growth factor binding protein (IGFBP-1), is significantly reduced after the exercise intervention. Physical activity has been shown to improve the symptom of fatigue.

The type, intensity, intensity and duration of the exercise to be applied differ from person to person. Exercise intervention is safe both during and after systemic treatments. Therefore, exercise intervention should be prescribed to breast cancer patients and they should be encouraged to maintain their established exercise habits or adopt a correct type of exercise.

The most widely accepted exercise regimen for breast cancer patients is about 150 minutes of moderate to vigorous intensity aerobic exercise per week. However, only 30% to 47% of breast cancer survivors are reported to adhere to the recommended exercise programs. Furthermore, aerobic exercise, strengthening exercises or body-mind exercises have a significant impact on side effects after cancer treatments. Aerobic and resistance exercises reduce physical and psychosocial problems associated with cancer and cancer treatment. Breast cancer survivors are also recommended mindfulness, yoga or body-mind exercises to feel better and more relaxed. Breathing exercises during physical activity are important for relaxation.

The 6-minute walk test (6MWD) is a widely used test for indirect measurement of cardiorespiratory fitness in various cancer populations. Studies have proven that the 6MWT is safe and feasible in breast cancer patients. The concept of 'can do, do do' has recently emerged to describe impaired physical functions in chronic obstructive pulmonary disease (COPD) and asthma. This concept categorizes investigators into four quadrants based on physical activity level and functional capacity measurements and cut-off point. This concept has proven useful for measuring physical function in both asthma and COPD. This concept may be useful in understanding physical functioning in breast cancer patients. Therefore, The aim of this study is to apply the concept of 'can do, do do' in breast cancer patients, to determine the quadrants according to physical activity level and functional capacity measurements in breast cancer patients, to investigate whether and to what extent there is a difference, whether and to what extent there is a difference between demographic information, disease stages, comorbidity level, clinical features, peripheral muscle strength, fatigue and quality of life and upper extremity functionality according to quadrants.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 18-65 years of age,
2. Volunteering to participate in the research,
3. At least 15 months after breast cancer surgery,
4. Six months after active breast cancer treatment (i.e. surgery/chemotherapy),
5. No problems in reading and/or understanding the scales and being able to cooperate with the tests,

Exclusion Criteria:

1. Presence of active infection,
2. Musculoskeletal and neurological diseases that may affect exercise performance, symptomatic heart disease,
3. Have a neurological disease or other clinical diagnosis that may affect cognitive status.
4. Musculoskeletal and neurologic disease, symptomatic heart disease, previous lung surgery and malignant disease that may affect exercise performance.
5. Presence of unstable hypertension or diabetes mellitus

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65 who were diagnosed with breast cancer in Hacettepe University Hospital, Department of Internal Medicine, Department of Medical Oncology and volunteered to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Functional Exercise Capacity | One Year
  Six-minute walk test (6MWT)
Physical Activity Level | One Year
  SenseWear Armband (SWA)

SECONDARY OUTCOMES:
Comorbidity Assessment | One Year
  The Charlson Comorbidity Index According to this index developed by the Institute of Medicine, comorbid diseases are assessed according to their severity. is scored. Comorbidities are scored from mild disease state to severe disease state. are given a score of 1, 2, 3, 4, respectively, and the score obtained by summing the scores of comorbid diseases The severity of comorbidity is also calculated according to the weighted score. One point for every ten years over the age of forty (50-59: 1 point, 60-69: 2 points, etc.)
Peripheral muscle strength assessment | One Year
  Peripheral muscle strength (knee extensors, shoulder abductors and hand grip strength) will be measured using a handheld digital dynamometer
Evaluation of Upper Extremity Functionality | One Year
  Questionnaire Disability of Arm, Shoulder and Hand (Q-DASH) Each item is scored on a 5-point Likert scale (1-5).The maximum score is 100 points. Score increase shows an increase in disability
Fatigue Assessment | One Year
  Piper Fatigue Scale (PFS) Responses for each item It is evaluated between 0-10 points. The total fatigue score is based on 22 items scores are summed and divided by the number of items. Scale obtained from high scores indicate a high level of perceived fatigue shows.
Evaluation of Quality of Life | One Year
  European Organization for Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) All scores were linearly transformed to a 0 to 100 scale. A high or healthy level of functioning is represented by a high functional score

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Calik-Kutukcu, PhD, Principal Investigator — Hacettepe University; Melda Saglam, PhD, Study Chair — Hacettepe University
Locations (1):
- Ebru Çalık Kutukcu, Ankara, Hacettepe Unıversity, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No